CLINICAL TRIAL: NCT05105555
Title: The e-BILD Study: Effects of Electric Nicotine Delivery Systems (ENDS) on Pulmonary Health in Teenagers.
Brief Title: The e-BILD Study: Effects of E-cigarettes on Lung Health in Teenagers.
Acronym: e-BILD
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: YTCR3419
Record Dates: First submitted 2021-09-20; First posted 2021-11-03 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Vaping; Lung Diseases
MeSH Terms: conditions — Vaping; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, Saliva, Nasal epithelial cells (obtained by nasal brushing)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: In this study, participants of the Bern Basel Infant Lung Development (BILD) cohort, a birth cohort of healthy term-born infants and their follow-up, will serve as healthy, non-vaping controls.
- Vaping teenagers: Vaping teenagers will be recruited independently from the BILD study through advertisements and visits to Bernese schools.

SUMMARY:
Electronic nicotine delivery systems (ENDS/e-cigarettes/vaping) are increasingly popular among teenagers around the world. The safety and potential adverse effects of ENDS in this population are largely unknown. While the aerosol, that users inhale, appears safe under laboratory conditions, there are still open questions, which have not yet been assessed. These cover (a) differences in exposure to chemicals (such as metabolites of Volatile Organic Compounds (VOCs) and metabolites of Polycyclic Aromatic Hydrocarbons (PAHs)) between healthy teenagers using ENDS and healthy teenagers not vaping, (b) effects of exposure to such chemicals on the body (measured by lung health indicators: airway symptoms such as coughing; lung function and lung structure tests; immune response of airway cells exposed to vapor; markers of oxidative stress), and (c) the role of nicotine metabolism. It is unknown which lung health indicator/s is/are most relevant to assess the effect of ENDS on lung health in teenagers.

The primary hypothesis of this study is that there will be differences in exposure to chemicals, resulting in more or more severe airway symptoms in vaping teenagers compared to their non-vaping peers. While there might not yet exist any differences regarding lung function or structure, we expect already visible effects of vaping on the local immune response of primary cells isolated from airways in vaping teenagers as compared to non-vaping peers.

In this study, participants of the Bern Basel Infant Lung Development (BILD) cohort, a birth cohort of healthy term-born infants and their follow-up, will serve as healthy, non-vaping controls.1 Vaping teenagers will be recruited independently from the BILD study through advertisements and visits to Bernese schools. Both populations combined represent the study population of the e-BILD study. All e-BILD study participants will undergo the same investigations. While these are currently planned for once in a time (so-called cross-sectional design) to compare results from non-vaping BILD study participants to otherwise healthy but vaping teenagers, repeated measures might follow, depending on the findings of the first phase.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* BILD study participants: see inclusion criteria of BILD study (NCT04286464), non-vaping
* e-BILD: healthy, term-born, vaping at least weekly (might include healthy, vaping participants from BILD)

Exclusion Criteria:

• None, except for general exclusion criteria of BILD study (NCT04286464)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In this study, participants of the Bern Basel Infant Lung Development (BILD) cohort, a birth cohort of healthy term-born infants and their follow-up, will serve as healthy, non-vaping controls. Vaping teenagers will be recruited independently from the BILD study through advertisements and visits to Bernese schools. Both populations combined represent the study population of the e-BILD study. All e-BILD study participants will undergo the same investigations. While these are currently planned for once in a time (so-called cross-sectional design) to compare results from non-vaping BILD study participants to otherwise healthy but vaping teenagers, repeated measures might follow, depending on the findings of the first phase.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Correlation of the respiratory symptom coughing with vaping status (validated by exposure markers) | At baseline
  Questions on frequency and intensity of coughing in past 12 months.
  Assessment of exposure markers (urinary concentrations of metabolites of VOCs (volatile organic compounds), urinary concentrations of metabolites of PAHs (Polycyclic aromatic hydrocarbons), urinary concentrations of urinary TSNA (Tobacco Specific Nitrosamines), urinary concentration of nicotine metabolites) to discriminate between vapers and non-vapers [Time Frame: at baseline]
  Urine sampling
Correlation of the respiratory symptom wheezing with vaping status (validated by exposure markers) | At baseline
  Questions on frequency and intensity of wheezing in past 12 months.
  Assessment of exposure markers (urinary concentrations of metabolites of VOCs (volatile organic compounds), urinary concentrations of metabolites of PAHs (Polycyclic aromatic hydrocarbons), urinary concentrations of urinary TSNA (Tobacco Specific Nitrosamines), urinary concentration of nicotine metabolites) to discriminate between vapers and non-vapers [Time Frame: at baseline]
  Urine sampling

SECONDARY OUTCOMES:
Correlation of validated vaping status with lung function (spirometry) in healthy teenagers | At baseline
  Assessment of lung function (spirometry)
Correlation of validated vaping status with lung function (bodyplethysmography) in healthy teenagers | At baseline
  Assessment of lung function (bodyplethysmography)
Correlation of lung function (multiple breath washout) in healthy teenagers | At baseline
  Assessment of lung function (multiple breath washout)
Correlation of validated vaping status with airway inflammation (exhaled nitric oxide) in healthy teenagers. | At baseline
  Assessment of levels of exhaled nitric oxide (eNO) measured by chemoluminescence analyzers in combination with ultrasound-based flow measurement.
Correlation of validated vaping status with lung structure (magnetic resonance imaging, MRI) in healthy teenagers. | At baseline
  Assessment of regional lung perfusion and ventilation.
Correlation of validated vaping status with measures of oxidative stress in healthy teenagers. | At baseline
  Measurement of oxidative stress metabolites in urine.
Correlation of validated vaping status with ex vivo immune response of nasal epithelial cells in healthy teenagers. | At baseline
  Assessment of nasal epithelial cell immune response collected by nasal brushing.
Role of nicotine metabolism on lung health indicators. | At baseline
  Measurement of nicotine metabolites in urine and saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Jakob, MD, Principal Investigator — Institute of Primary Health Care BIHAM, Bern University; Reto Auer, MD, MAS, Principal Investigator — Institute of Primary Health Care BIHAM, Bern University; Philipp Latzin, MD, PhD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Insel, Bern University Hospital, Bern, Switzerland